CLINICAL TRIAL: NCT01752322
Title: Efficacy and Safety of Lidocaine 5% Medicated Plaster in Localized Chronic Post-operative Neuropathic Pain
Brief Title: Efficacy and Tolerability of Lidocaine Plaster for Treatment of Long-term Local Nerve Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KF10004/10; 2012-000347-28 (EudraCT Number)
Record Dates: First submitted 2012-09-12; First posted 2012-12-19 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Pain; Chronic Pain; Neuropathic Pain; Postoperative Pain
MeSH Terms: conditions — Pain; Chronic Pain; Neuralgia; Pain, Postoperative | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine plaster (Experimental): Topical hydrogel plaster
  Interventions: Drug: Lidocaine 5% medicated plaster
- Placebo plaster (Placebo Comparator): Topical hydrogel plaster
  Interventions: Drug: Placebo plaster

INTERVENTIONS:
Drug: Lidocaine 5% medicated plaster
  Arms: Lidocaine plaster
Drug: Placebo plaster
  Arms: Placebo plaster

SUMMARY:
The purpose of this trial is to investigate the efficacy and safety of lidocaine 5% medicated plaster in localized chronic post-operative neuropathic pain in comparison to placebo plaster.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years or older.
* Subjects suffering from moderate to severe localized chronic PoNP (post operative neuropathic pain) pain following surgery (e.g., thoracotomy, total/partial knee replacement, cholecystectomy, mastectomy, inguinal hernia repair, varicose vein stripping).
* Localized PoNP present for at least 3 months.
* Size of the affected painful skin area is not larger than the size of 3 plasters.
* Intact skin besides the scar of surgery in the area of plasters application
* Baseline average pain intensity of 4 or greater on the 11 point pain intensity Numeric Rating Scale.

Exclusion Criteria:

* Participation in another trial (with medicine or a device under investigation) in parallel or less than 30 days prior to enrollment in this trial.
* Previous enrollment in this trial.
* History of dependency or active drug abuse (alcohol, medication) during the 1 year prior to enrollment.
* Evidence or history (during the 3 years prior to enrollment) of neurotic personality or psychiatric illness that in the investigator's opinion may affect efficacy or safety assessments or may compromise the subjects safety during trial participation.
* Pregnant or breastfeeding women or women of childbearing potential who are sexually active without satisfactory contraception.
* Any surgery performed in the 3 months prior to enrollment, which may affect efficacy or safety assessment.
* Any surgery scheduled or expected during the trial.
* Clinically significant disease (e.g., acquired immunodeficiency syndrome) or condition that may affect efficacy or safety assessments, or any other reason which, in investigator's opinion, may preclude the subject's participation in the trial.
* History of malignancy (with the exception of neoplasia related to the trial indication) within 2 years prior to enrollment.
* Subject with PoNP related to a surgery due to neoplasia: suspected residual neoplasia or metastases.
* Pending litigation due to chronic pain or disability.
* Total anesthesia in the cutaneous area neurologically related to the location of the surgical intervention.
* Hypersensitivity to the lidocaine 5% medicated plaster, its excipients, or anesthetics of the amide type.
* Any former use of topical lidocaine in the area of localized chronic PoNP.
* Severe renal, hepatic or heart disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline of recorded average pain intensity values during the last 24 hours, averaged over the 7 days of Week 12 of the Double-blind Treatment Period. | Days 78-85

SECONDARY OUTCOMES:
Mean pain intensity based on the average pain intensity during the last 24 hours, calculated over the last 4 weeks and 12 weeks of the Double blind Treatment Period. | up to 12 weeks
Mean pain intensity based on the current pain intensity before plaster removal, calculated over the last 7 days, 4 weeks, and 12 weeks of the Double blind Treatment Period. | up to 12 weeks
Weekly mean pain intensity before plaster removal based on the average pain intensity during the last 24 hours. | up to 12 weeks
Weekly mean pain intensity before plaster removal based on current pain intensity before plaster removal. | up to 12 weeks
Final score of the painDETECT Pain Questionnaire during the Double blind Treatment Period. | Day 85
Pain intensity from mechanical dynamic allodynia (brush) testing. | Day 85
Anxiety and depression scores of HADS. | Day 85
The weighted Health Status Index of quality of life by means of EQ 5D. | Day 85
Total score in quality of sleep using CPSI. | Day 85
Mean pain intensity change from baseline based on the average pain intensity during the last 24 hours, calculated over the last 4 weeks and 12 weeks of the Double blind Treatment Period. | up to 12 weeks
Mean pain intensity change from baseline based on the current pain intensity before plaster removal, calculated over the last 7 days, 4 weeks, and 12 weeks of the Double blind Treatment Period. | up to 12 weeks
Weekly mean pain intensity change from baseline before plaster removal based on the average pain intensity during the last 24 hours. | up to 12 weeks
Weekly mean pain intensity change from baseline before plaster removal based on current pain intensity before plaster removal. | up to 12 weeks
Change from baseline in the total score of the painDETECT Pain Questionnaire during the Double blind Treatment Period. | Day 85
Change from baseline in pain intensity from mechanical dynamic allodynia (brush) testing. | Day 85
Change from baseline in anxiety and depression scores of HADS. | Day 85
Change from baseline in total score of quality of life by means of EQ 5D. | Day 85
Change from baseline in total score in quality of sleep using CPSI. | Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Grünenthal GmbH
Locations (42):
- Austria (6):
  - AUT004, Klagenfurt
  - AUT005, Senftenberg
  - AUT001, Vienna
  - AUT006, Vienna
  - AUT002, Vienna
  - AUT003, Vienna
- Belgium (5):
  - BEL001, Gozée
  - BEL006, Halen
  - BEL004, Ham
  - BEL007, Lanaken
  - BEL002, Natoye
- Brazil (7):
  - BRA005, Barretos
  - BRA002, Itajaí
  - BRA001, Porto Alegre
  - BR008, Salvador
  - BRA003, São Paulo
  - BRA006, São Paulo
  - BRA007, São Paulo
- Denmark (3):
  - DNK005, Copenhagen
  - DNK004, Glostrup Municipality
  - DNK001, Odense
- France (10):
  - FRA004, Amiens
  - FRA002, Bordeaux
  - FRA001, Boulogne-Billancourt
  - FRA003, Le Chesnay
  - FRA005, Lille
  - FRA010, Montauban
  - FRA006, Nantes
  - FRA009, Paris
  - FRA008, Saint-Priest-en-Jarez
  - FR007, Toulouse
- Italy (3):
  - ITA004, Florence
  - ITA003, Napoli
  - ITA001, Rome
- Spain (4):
  - ESP001, Barcelona
  - ESP002, Barcelona
  - ESP006, Madrid
  - ESP005, Madrid
- United Kingdom (4):
  - GBR003, Cardiff
  - GBR001, Glasgow
  - GBR004, Liverpool
  - GBR002, Manchester

REFERENCES:
- [Derived] Palladini M, Boesl I, Koenig S, Buchheister B, Attal N. Lidocaine medicated plaster, an additional potential treatment option for localized post-surgical neuropathic pain: efficacy and safety results of a randomized, placebo-controlled trial. Curr Med Res Opin. 2019 May;35(5):757-766. doi: 10.1080/03007995.2019.1565709. Epub 2019 Jan 21. PMID 30614286